CLINICAL TRIAL: NCT05888363
Title: Complications in the Management and Removal of Rectal and Vaginal Foreign Bodies
Brief Title: Management and Removal of Foreign Bodies in the Emergency Department
Status: Completed | Type: Observational
Sponsor: Arrowhead Regional Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 20-46a
Record Dates: First submitted 2023-05-24; First posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2021-12

CONDITIONS: Rectal Foreign Body; Rectal Perforation; Colonic Perforation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Rectal foreign body removed in emergency department: All patients where the removal of the rectal foreign body was successful in the emergency department
  Interventions: Other: No Intervention
- Rectal foreign body removed in operating room: All patients where the removal of the rectal foreign body was not successful in the emergency department and required removal in the operating room
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — Difference in outcomes in patients with rectal foreign bodies removed in the emergency department or in the operating room.

SUMMARY:
Management of rectal foreign bodies presents unique challenges in the emergency department. Rectal foreign bodies may consist of various compositional materials and ergonomics which include but are not limited to vegetables, light bulbs, everyday household items, and body packing of illicit drugs. Patients presenting to the emergency department with rectal foreign bodies range widely in age from prepubertal patients to older adults. Insertion of rectal foreign bodies have been classified as voluntary or involuntary, as well as sexual or non-sexual. The definition of rectal foreign bodies can be blurry, as many objects inserted via the rectum are large enough to enter the sigmoid colon. Although detailed epidemiologic data are scant, recent studies reported a progressive rise in complications related to rectal foreign bodies with incidence disproportionately higher in men and an average age in the mid 40s.

DETAILED DESCRIPTION:
rectal foreign bodies have been reported to result in a varying range of complications. According to the Rectal Organ Injury Scale (ROIS) proposed by the American Association for the Surgery of Trauma, injuries caused by rectal foreign bodies range from Grade I to Grade V. Grade I injury is defined as hematoma without devascularization. Grade II injury includes partial thickness laceration less than 50% of circumference while Grade III injury demonstrates partial thickness laceration greater than 50% of circumference. Grade IV injury is noted as a full-thickness laceration extending into the perineum. Grade V injury demonstrates devascularized segment. Colonic organ injury scale grading is very similar to the ROIS with differences consisting of transection of the colon in grade IV and transection of the colon with devascularized segment and tissue loss in grade V. Prior studies suggest that most injuries resulting from inserted objects are classified as Grade I injuries.

Investigators from two separate studies suggested a nearly 10% complication rate in cases of attempted transanal bedside removals in the ED. The most commonly reported complications of bedside procedures were perforation of the rectum, followed by the rectal mucosal injury. One particular study noted that 17% of patients sustained perforation of colon. The underlying cause for such high rates of complications may be multifactorial, including the status of the patients, the presence of comorbidities, and delays in presentation to the hospital. To reduce the rate of complication various extraction methods such as the use of sigmoidoscopy. With the increased incidence of rectal foreign bodies and the associated complications, it is imperative to explore and determine a set of standards for the safe and effective removal of rectal foreign bodies. However, current literature is not clear as to the ideal setting. This study aims to further explore various methods of extraction, outcomes and complications associated with bedside attempts at removal of rectal foreign bodies.

ELIGIBILITY:
Inclusion Criteria:

* Rectal foreign body removal
* Colonic foreign body removal
* Vaginal foreign body removal
* Foreign body removals performed in the emergency department

Exclusion Criteria:

* All individuals under the age of 18

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: To evaluate the safety of foreign body removals in the emergency department and in the operating room in patients older than 18 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2021-12-08 (Actual); Study Completion 2021-12-08 (Actual)

PRIMARY OUTCOMES:
Surgical site infections within the first 30 days | 30 days
  Infection along surgical incision
Length of Hospital Stay | 360 days
  Length of total hospital stay from admission in the hospital
Hospital Mortality | 30 days
  Survival within the first 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Michael M Neeki, DO, Principal Investigator — Arrowhead Regional Medical Center
Locations (1):
- Arrowhead Regional Medical Center, Colton, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ooi BS, Ho YH, Eu KW, Nyam D, Leong A, Seow-Choen F. Management of anorectal foreign bodies: a cause of obscure anal pain. Aust N Z J Surg. 1998 Dec;68(12):852-5. doi: 10.1046/j.1440-1622.1998.01463.x. PMID 9885867
- [Background] Sei H, Tomita T, Nakai K, Nakamura K, Tamura A, Ohda Y, Oshima T, Fukui H, Watari J, Miwa H. Rectal Foreign Body of Eggplant Treated Successfully by Endoscopic Transanal Removal. Case Rep Gastroenterol. 2018 Apr 26;12(1):189-193. doi: 10.1159/000488974. eCollection 2018 Jan-Apr. PMID 29805365
- [Background] Traub SJ, Hoffman RS, Nelson LS. Body packing--the internal concealment of illicit drugs. N Engl J Med. 2003 Dec 25;349(26):2519-26. doi: 10.1056/NEJMra022719. No abstract available. PMID 14695412
- [Background] Rodriguez-Hermosa JI, Codina-Cazador A, Ruiz B, Sirvent JM, Roig J, Farres R. Management of foreign bodies in the rectum. Colorectal Dis. 2007 Jul;9(6):543-8. doi: 10.1111/j.1463-1318.2006.01184.x. PMID 17573750